CLINICAL TRIAL: NCT05523492
Title: Pathways and Barriers to Access and Utilization of Internet-Delivered Cognitive Behaviour Therapy (ICBT) by Diverse Ethnocultural People of Saskatchewan
Brief Title: Exploring Use of Internet-Delivered Cognitive Behaviour Therapy (ICBT) by Diverse Ethnocultural People of Saskatchewan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Regina (Other)
Collaborators: Saskatchewan Health Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-197b
Record Dates: First submitted 2022-08-29; First posted 2022-08-31 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Anxiety; Depression
Keywords: anxiety; depression; therapist-assistance; internet-delivered cognitive behaviour therapy; patient-centred therapy; knowledge implementation; mental health system
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Culturally Enhanced Wellbeing Course (Experimental): For this study, the ICBT program, called the Wellbeing Course was culturally enhanced by simplifying language for individuals with limited command of English, acknowledging cultural differences and increase representation in imagery. Audiovisual components were included to provide a brief summary of each lesson. Furthermore, additional client stories were added to the intervention to diversify narratives and be more representative of the clients seeking this intervention.
  Interventions: Behavioral: Internet-delivered Cognitive Behavioural Therapy

INTERVENTIONS:
Behavioral: Internet-delivered Cognitive Behavioural Therapy — All clients will receive the Culturally Enhanced Wellbeing Course. The Course was originally developed at Macquarie University in Australia and was then culturally enhanced by the Online Therapy Unit in Saskatchewan Canada. The course is a trans-diagnostic Internet-delivered cognitive behaviour therapy intervention targeting symptoms of depression and anxiety. It comprises 5 online lessons targeting: 1) symptom identification and the cognitive behavioural model; 2) thought monitoring and challenging; 3) de-arousal strategies and pleasant activity scheduling; 4) graduated exposure; and 5) relapse prevention. Materials are presented in a didactic (i.e., text-based with visual images) and case-enhanced learning format (i.e., educational stories demonstrate the application of skills) and include homework activities. Lessons are released gradually in order over 8 weeks. Therapists will spend ~15 mins. per week/per client offering support via emails and or phone calls.

SUMMARY:
In an attempt to increase timely and accessible psychological treatment for depression and anxiety, Internet-delivered Cognitive Behaviour Therapy (ICBT) has emerged. In ICBT, patients review treatment materials online and complete relevant exercises to learn cognitive behavioural strategies. They also commonly access brief therapist support through weekly emails or phone calls.

Data analysis of ICBT offered via the Online Therapy Unit in Saskatchewan has found lower participation in ICBT among individuals from diverse (non-white/ Caucasian) ethnocultural backgrounds. Furthermore, feedback from participants has identified opportunities to improve ICBT by: 1) simplifying language to improve clarity; 2) adding audiovisual content to aid with learning ICBT strategies; and 3) adding in diverse examples/stories to show applicability of ICBT to individuals with diverse backgrounds. The purpose of this study is to evaluate an ICBT program that has been improved in this way, called the Culturally Enhanced Wellbeing Course. Specifically, the observational pilot study with 30 clients from diverse ethnocultural backgrounds aims to examine improvements in depression and anxiety from pre to post treatment as well as patient experiences with the Culturally Enhanced Wellbeing Course.

DETAILED DESCRIPTION:
In the last 10 years, the Online Therapy Unit has successfully provided ICBT to more than 10000 people experiencing mental health problems and there has been a growing demand and utilization of ICBT in Saskatchewan. However, a recent analysis of service utilization trends over six years shows that there has been a consistently low (11%) participation from the people of diverse (non-white/ Caucasian) ethnocultural groups in the ICBT program, called the Wellbeing Course. Furthermore, the number of ICBT lessons completed by the participants of diverse ethnocultural backgrounds was significantly lower compared to white/Caucasian participants.

Review of feedback from participants from diverse ethnocultural backgrounds indicated a need to simplify the language of the course, and diversify the narratives in the stories which accompany the lessons to illustrate how the exercises can be used and how past participants have found the course. Participants also suggested the addition of audiovisual elements in conjunction with text throughout the lessons to improve understanding of materials.

In this study, we will aim to evaluate the Culturally Enhanced Wellbeing Course among 30 treatment-seeking adults in Saskatchewan from diverse cultural backgrounds.

The Culturally Enhanced Wellbeing Course will be evaluated through pre-post-treatment assessments using self-report questionnaires and individual semi-structured telephone interviews conducted toward the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Endorse symptoms of anxiety or depression
* Resident of Saskatchewan
* Access to a computer and the Internet
* Self-identifying as having a diverse ethnocultural background

Exclusion Criteria:

* Have a severe unmanaged psychiatric illness (e.g. psychosis)
* Assessed as being at high risk of suicide
* Report severe problems with alcohol or drugs
* Report severe cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2022-06-14 (Actual); Primary Completion 2023-02-20 (Actual); Study Completion 2023-02-20 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire 9-item (PHQ-9) | Baseline (Screening), weeks 1-8, and 20 week from enrollment
  Tracking the change in depression symptoms. 9 items are summed into a total score, with scores ranging from 0 to 27. Higher scores are associated with higher depression severity.
Generalized Anxiety Disorder 7-item (GAD-7) | Baseline (Screening), weeks 1-8 and 20 week from enrollment
  Tracking the change in anxiety symptoms. 7 items are summed into a total score ranging from 0 to 21, with higher scores indicating more severe self-reported levels of anxiety.
ICBT Experience Interview Guide | Week 6
  This measure includes 12 items to gain feedback on participant experience of Wellbeing Course.
Mid-point Additional Resource Satisfaction Questionnaire | Week 4 from enrollment
  Gathering feedback on the Additional Resources up to this time point. This measure includes 3 questions, one in which is open-ended.
Post-treatment Additional Resource Satisfaction Questionnaire | Week 8 from enrollment
  Gathering feedback on the Additional Resources up to this time point. This measure includes 3 questions, one in which is open-ended.
Mid-point Patient Story Satisfaction Questionnaire | Week 4 from enrollment
  Gathering feedback on the patient stories up to this time point. This measure includes 4 questions to quantify quality of participant Stories.
Post-treatment Patient Story Satisfaction Questionnaire | Week 8 from enrollment
  Gathering feedback on the patient stories up to this time point. This measure includes 4 questions to quantify quality of participant Stories.

SECONDARY OUTCOMES:
Adjustment Disorder New Model 8 (ADNM) | Baseline (Screening) week 8 and week 20 from enrollment
  Measure includes 8 questions to determine severity of impact of a specific event. High scores indicate a greater degree of Adjustment Disorder
Treatment Satisfaction | Week 8 from enrollment
  Measure includes 17 questions assessing satisfaction with various aspects of ICBT and also negative effects of treatment. Items are not summed but are examined individually.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Hadjistavropoulos, PhD, Principal Investigator — University of Regina
Locations (1):
- Department of Psychology, Regina, Saskatchewan, Canada

REFERENCES:
- [Derived] Sapkota RP, Valli E, Dear BF, Titov N, Hadjistavropoulos HD. Satisfaction, engagement, and outcomes in internet-delivered cognitive behaviour therapy adapted for people of diverse ethnocultural groups: an observational trial with benchmarking. Front Psychiatry. 2024 Mar 4;15:1270543. doi: 10.3389/fpsyt.2024.1270543. eCollection 2024. PMID 38501087